CLINICAL TRIAL: NCT06532604
Title: Study of Electrophysiological Markers of Antidepressants in Major Depressive Disorder
Acronym: MESANTIDEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00551-46; RIPH 2024-01 (Other: Centre Psychothérapique de Nancy)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Antidepressant; Electroretinography; Precision psychiatry; Selective Serotonin Reuptake Inhibitor; Alpha-2 adrenergic receptor antagonists; Retinal function
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroretinography

STUDY DESIGN:
Intervention Model Description: MESANTIDEP is a pilot, longitudinal, prospective and multicenter cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSRI treated patients (Experimental): MDD patients treated with Selective Serotonin Reuptake Inhibitors (SSRIs) the day after the inclusion visit.
  Interventions: Device: Electroretinography (ERG)
- Alpha-2 antagonists treated patients (Experimental): MDD patients treated with alpha-2 adrenergic receptor antagonists (alpha-2 antagonists) the day after the inclusion visit.
  Interventions: Device: Electroretinography (ERG)

INTERVENTIONS:
Device: Electroretinography (ERG) — ERG are specifically carried out for research. They are performed in Nancy with the MonPackOne device developed by Metrovision for participants at center n°1, and in Paris with the RETeval device developed by LKS Technologie for participants at center n°2. Both devices comply with ISCEV standard and are CE marked. They enable the reccord of Pattern ERG, Flash ERG and Multifocal ERG using corneal and skin electrodes, or Sensor Strip skin electrodes only, for the Nancy and Paris centers respectively.
  Other Names: MonPackOneⓇ (Métrovision); RETevalⓇ (LKS technologie)

SUMMARY:
Major depressive disorder (MDD) is a frequent and particularly disabling disorder. The efficacy of current antidepressants is limited, with 50-60% of patients not achieving a sufficient response to treatment. Indeed, to date, clinicians are unable to predict the therapeutic response a patient will obtain to a given molecule. This often results in several trials of a molecule until clinical efficacy is achieved, with a delay of several months of untreated disease. Achieving faster efficacy by targeting the right molecule for each patient in the 1st line of treatment would limit the morbidity and mortality induced by MDD, and its impact on quality of life. To achieve this goal rapidly, there is a need to identify markers for predicting and monitoring therapeutic response to antidepressants.

This is why the MESANTIDEP study aims to propose electroretinographic (ERG) biomarkers for predicting therapeutic response at 12 weeks for the two main therapeutic classes of antidepressants prescribed as 1st-line treatment for major depressive disorder: Selective Serotonin Reuptake Inhibitors (SSRIs) and alpha-2 adrenergic receptor antagonists (alpha-2 antagonists). Secondly, investigators will look for ERG biomarkers of therapeutic response at 6 weeks, and 12 weeks, for these two therapeutic classes of antidepressants.

For this purpose, patients diagnosed with MDD and requiring the initiation of an antidepressant - of the SSRI or alpha-2-antagonist class - will be included. At their inclusion visit, patients will not yet have started their antidepressant treatment and will undergo various tests. These include clinical questionnaires, sleep assessment questionnaires and three ERG tests (fERG, PERG and mfERG). Antidepressant treatment can be started by the patient the day after the inclusion visit. 6 and 12 weeks later, the patient undergoes the same tests as at the inclusion visit to monitor their therapeutic response to the prescribed antidepressant. The identification of electrophysiological markers predictive of therapeutic response to antidepressants is intended to help clinicians in the treatment of MDD patients. More rapid therapeutic intervention tailored to each patient will limit the functional impact, improve quality of life and reduce the morbidity and mortality associated with the disease. These electrophysiological ERG measurements are easy to perform. They are therefore accessible to all, and can be used, through a multimodal approach, in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a current unipolar depressive episode according to DSM-V criteria
* Prescription of antidepressant treatment - SSRI or alpha-2 antagonist - by the psychiatrist or referring physician for the current depressive episode
* Age 18 or more
* Affiliation with a welfare scheme and native French speakers
* Complete information on the study received and written informed consent signed

Exclusion Criteria:

* Diagnosis of a progressive psychiatric disorder (except MDD and anxiety disorder) according to DSM-V criteria
* Seasonal character of the depression
* Current antidepressant treatment
* Recommended antidepressant treatment other than SSRI or alpha-2 antagonist
* High suicide risk
* Retinal or ophtalmologic pathology affecting visual acuity as assessed by the Monoyer scale.
* History of head trauma, epilepsy or other neurological disorders
* Participation in another interventional study (including exclusion period)
* Intellectual disability leading to difficulty participating or impossibility or inability to understand the information provided on the study.
* Persons cited in Articles L. 1121-5 to L. 1121-8 of the French Public Health Code: pregnant women, parturient or breastfeeding mothers, persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care under duress, persons admitted to a health or social establishment for other goals than research, minors, adults subject to a legal protection, adults who are unable to express their consent and who are not subject to a legal protection measure.
* Criteria incompatible with the use of the ERG device: open wound in an area covered or enveloped by the device; implantable medical device (e.g. pacemaker); user at high risk of contagion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
ERG amplitudes at baseline | Baseline (D0)
  Modification of amplitude measured with flash, pattern and multifocal electroretinogram amplitude in microvolt
ERG implicit times at baseline | Baseline (D0)
  Modification of implicit time measured with flash, pattern and multifocal electroretinogram implicit time in millisecond
Montgomery Asberg Depression Rating Scale score differences between D0 and W12 | Baseline (D0) and 12 weeks after baseline (W12)
  A subject will be declared responder (decrease greater than or equal to 8 points between D0 and W12) or non-responder (score difference less than 8 points or increase between D0 and W12). We obtain binary data (responder/non-responder).

SECONDARY OUTCOMES:
ERG amplitudes | Baseline (D0)
  Modification of amplitude measured with flash, pattern and multifocal electroretinogram amplitude in microvolt
ERG amplitudes | 6 weeks after baseline (W6)
  Modification of amplitude measured with flash, pattern and multifocal electroretinogram amplitude in microvolt
ERG amplitudes | 12 weeks after baseline (W12)
  Modification of amplitude measured with flash, pattern and multifocal electroretinogram amplitude in microvolt
ERG implicit time | Baseline (D0)
  Modification of implicit time measured with flash, pattern and multifocal electroretinogram implicit time in millisecond
ERG implicit time | 6 weeks after baseline (W6)
  Modification of implicit time measured with flash, pattern and multifocal electroretinogram implicit time in millisecond
ERG implicit time | 12 weeks after baseline (W12)
  Modification of implicit time measured with flash, pattern and multifocal electroretinogram implicit time in millisecond
Montgomery Asberg Depression Rating Scale (MADRS) score differences | Baseline (D0) and 12 weeks after baseline (W12)
  A subject will be declared responder (decrease greater than or equal to 8 points between D0 and W12) or non-responder (score difference less than 8 points or increase between D0 and W12). We obtain binary data (responder/non-responder).
Montgomery Asberg Depression Rating Scale (MADRS) score differences | Baseline (D0) and 6 weeks after baseline (W6)
  Differences in MADRS scores
Montgomery Asberg Depression Rating Scale (MADRS) score differences | 6 weeks after baseline (W6) and 12 weeks after baseline (W12)
  Differences in MADRS scores

OTHER OUTCOMES:
Alcohol Use DIsorders Test (AUDIT) | Baseline (D0)
  A questionnaire rating consumption of alcoholic drinks
Fagerström test | Baseline (D0)
  A questionnaire rating cigarette consumption
Montgomery-Asberg Depression Rating Scale (MADRS) self | Baseline (D0)
  An auto-rating scale measuring depressive symptoms
Montgomery-Asberg Depression Rating Scale (MADRS) self | 6 weeks after baseline (W6)
  An auto-rating scale measuring depressive symptoms
Montgomery-Asberg Depression Rating Scale (MADRS) self | 12 weeks after baseline (W12)
  An auto-rating scale measuring depressive symptoms
Hamilton Anxiety Rating Scale (HAM-A) | Baseline (D0)
  A questionnaire rating level of anxiety
Hamilton Anxiety Rating Scale (HAM-A) | 6 weeks after baseline (W6)
  A questionnaire rating level of anxiety
Hamilton Anxiety Rating Scale (HAM-A) | 12 weeks after baseline (W12)
  A questionnaire rating level of anxiety
Geriatric Depression Scale (GDS) | Baseline (D0)
  A questionnaire measuring depressive symptoms for patients over 65
Geriatric Depression Scale (GDS) | 6 weeks after baseline (W6)
  A questionnaire measuring depressive symptoms for patients over 65
Geriatric Depression Scale (GDS) | 12 weeks after baseline (W12)
  A questionnaire measuring depressive symptoms for patients over 65
Medication Adherence Report Scale (MARS) | Baseline (D0)
  A questionnaire assessing patients' adherence to antidepressants
Medication Adherence Report Scale (MARS) | 6 weeks after baseline (W6)
  A questionnaire assessing patients' adherence to antidepressants
Medication Adherence Report Scale (MARS) | 12 weeks after baseline (W12)
  A questionnaire assessing patients' adherence to antidepressants
Pittsburgh Sleep Quality Index (PSQI) | Baseline (D0)
  A questionnaire assessing the subjective quality of sleep during the past month
Pittsburgh Sleep Quality Index (PSQI) | 6 weeks after baseline (W6)
  A questionnaire assessing the subjective quality of sleep during the past month
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks after baseline (W12)
  A questionnaire assessing the subjective quality of sleep during the past month
Epworth sleepiness scale (ESS) | Baseline (D0)
  A questionnaire assessing the daytime sleepiness
Epworth sleepiness scale (ESS) | 6 weeks after baseline (W6)
  A questionnaire assessing the daytime sleepiness
Epworth sleepiness scale (ESS) | 12 weeks after baseline (W12)
  A questionnaire assessing the daytime sleepiness
Insomnia Severity Index (ISI) | Baseline (D0)
  A questionnaire assessing the severity of insomnia
Insomnia Severity Index (ISI) | 6 weeks after baseline (W6)
  A questionnaire assessing the severity of insomnia
Insomnia Severity Index (ISI) | 12 weeks after baseline (W12)
  A questionnaire assessing the severity of insomnia

CONTACTS AND LOCATIONS:
Overall Officials: Schwitzer Thomas, Pr, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Deus M, Petit C, Moulard M, Cosker E, Mellouki Bendimred N, Albuisson E, Maruani J, Geoffroy PA, Schwitzer T. Exploring the ElectroRetinoGraphy as a biomarker for predicting and monitoring therapeutic response to antidepressants in major depressive disorder: study protocol for the MESANTIDEP trial. Front Psychiatry. 2025 Apr 25;16:1501166. doi: 10.3389/fpsyt.2025.1501166. eCollection 2025. PMID 40352365